CLINICAL TRIAL: NCT04254367
Title: Empowering Patients With Long-term Impaired Work Ability to Participate in Health Related Decisions
Brief Title: Empowering Patients to Participate in Health Care Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Learn-to-Cope
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Rehabilitation
Keywords: health literacy; sense of coherence; empowerment; patient education as topic; health-related quality of life; coping strategies; bio-psycho-social model
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Intervention Model Description: The study design is a cluster randomized controlled study comparing the intervention in addition to treatment as usual (TAU) with TAU. Follow-up is performed with validated questionnaires after 3, 6 and 12 months. Primary outcome is net inactivity days (net days without employment or rehabilitation) and secondary outcome variables are the number of net and gross days with sick leave during the follow-up period, sense of coherence, health literacy, health-related quality of life, confidence in own problem solving ability, work ability and work satisfaction, social function and health habits, symptoms of depression, anxiety, and exhaustion as well as pain and catastrophization. Randomization will be performed at PCC level. Around 30 PCCs and 400 patients will be included in the study. The intervention consists of patient education with study circles meeting half a day per week for eight following weeks.
Who Masked: Investigator
Masking Description: Investigator blinded of randomization results when informing PCCs about the study and PCCs blinded when selecting patients to the study. The PCCs were instructed to select 20-25 patients following the study's inclusion and exclusion criteria and among these select 12-14 patients to ask first. The other selected patients were to be asked if the first patients did not agree to participate in the study. After selection the PCCs were informed about randomization results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - experimental TAU + intervention (Experimental): Patient education in study circles, aiming to empower patients to participate in health care and rehabilitation by increasing health literacy and sense of coherence. The study circles will meet half a day each week for eight following weeks.
  Interventions: Behavioral: Learn-to-Cope
- TAU - no intervention (No Intervention): Treatment as usual following local routines on each primary care center

INTERVENTIONS:
Behavioral: Learn-to-Cope — Patient education in study circles, aiming to empower patients to participate in health care and rehabilitation by increasing health literacy and sense of coherence. The study circles will meet half a day each week for eight following weeks.
  Arms: Intervention group - experimental TAU + intervention

SUMMARY:
The study aims to evaluate whether an intervention with patient education in study circles, aiming to empower patients to participate in health care an rehabilitation by increasing health literacy and sense of coherence, may have a causal effect on perceived health, ability and function as well as independence and quality of life for patients with long-term health-related disabilities and passive coping strategies.

DETAILED DESCRIPTION:
Chronic poor health and impaired work ability entails both personal suffering and considerable social costs. Poverty, homelessness, difficulties to handle complex issues, and maltreatment may affect health outcomes in the long run. Both sense of coherence (SOC) and the ability to understand health-related information (health literacy) influences personal coping strategies and thus the motivation to participate in health care and rehabilitation, which is known to have a positive impact on health outcome. The purpose of this study is to evaluate whether an intervention with patient education in study circles, aiming to empower patients to participate in health care and rehabilitation by increasing health literacy and sense of coherence, may have a causal effect on perceived health, ability and function as well as independence and quality of life for patients with long-term health-related disabilities and passive coping strategies. The study design is a cluster randomized controlled study comparing the intervention in addition to treatment as usual (TAU) with TAU. Follow-up is performed with validated questionnaires after 3, 6 and 12 months. Primary outcome is net inactivity days (net days without employment or rehabilitation) and secondary outcome variables are the number of net and gross days with sick leave during the follow-up period, sense of coherence, health literacy, health-related quality of life, confidence in own problem solving ability, work ability and work satisfaction, social function and health habits, symptoms of depression, anxiety, and exhaustion as well as pain and catastrophization. Randomization will be performed at Primary Care Center (PCC) level. Around 30 Primary Care Centers and 400 patients will be included in the study. The intervention consists of patient education with study circles meeting half a day per week for eight following weeks. The study is expected to show whether patient education in study circles aiming to increase health literacy and sense of coherence has a causal effect on perceived health, ability and function, independence and quality of life for patients with long-term health-related disabilities and passive coping strategies compared to TAU.

The research subjects will answer all questionnaires in a web based tool approved for storing research data, esMaker (Entergate AB) on their mobile phone, iPad or computer. Individual web links to the questionnaires will be distributed via e-mail. Research subject identity is replaced with individual codes in esMaker. The research assistant will be in charge of the CodeKey and responsible for distributing the web links and for reminding the research subjects to fill in the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Patients attending primary care centers included in the study.

* Aged 18-64 years
* Health-related impaired work ability > 60 net days last 6 months

Exclusion Criteria:• Acute crisis

* Serious mental disorder needing psychiatric specialist care
* Serious somatic disease a definite barrier to rehabilitation for a foreseeable future
* Cognitive impairment or not speaking /understanding Swedish

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Net days with sceduled activity | Change from base-line net days with scedulded activity at 6 months
  What is the effect of interactive patient education in supervised study groups on net days with scheduled activity in patients of working age with long-term health-related work impairment (measured as change in net days with work / scheduled work preparatory rehabilitation (unemployed) / scheduled work preparatory rehabilitation during sick leave (on sick leave) from baseline to 6 months after baseline).

SECONDARY OUTCOMES:
Net days with sceduled activity | Change from base-line net days with scedulded activity at 3 months
  What is the effect of interactive patient education in supervised study groups on net days with scheduled activity in patients of working age with long-term health-related work impairment (measured as change in net days with work / scheduled work preparatory rehabilitation (unemployed) / scheduled work preparatory rehabilitation during sick leave (on sick leave) from baseline to 3 months after baseline).
Net days with sceduled activity | Change from base-line net days with scedulded activity at 12 months
  What is the effect of interactive patient education in supervised study groups on net days with scheduled activity in patients of working age with long-term health-related work impairment (measured as change in net days with work / scheduled work preparatory rehabilitation (unemployed) / scheduled work preparatory rehabilitation during sick leave (on sick leave) from baseline to 12 months after baseline).
Health-related quality of life | Change from base-line scores EQ-5D at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' health-related quality of life (measured by change in scores in EQ-5D from baseline to 3 months after baseline). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health-related quality of life | Change from base-line scores EQ-5D at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' health-related quality of life (measured by change in scores in EQ-5D from baseline to 6 months after baseline). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health-related quality of life | Change from base-line scores EQ-5D at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' health-related quality of life (measured by change in scores in EQ-5D from baseline to 12 months after baseline). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Sense of coherence (SOC) | Change from base-line scores SOC-13 scale at 3 months
  What is the effect of interactive patient education in supervised study groups on the participants' sense of coherence (measured by changes in scores in SOC-13 scale in Swedish9 from baseline to 3 months after baseline). Antonovsky developed the 29 item Orientation to Life Questionnaire to measure the sense of coherence, having 11 items measuring comprehensibility, 10 items measuring manageability, and 8 items measuring meaningfulness. The response alternatives are a semantic scale of 1 point to 7 points. The questionnaire yields a summed score with a range from 29 to 203. A shorter version of 13 questions of the original form was developed by Antonovsky, where the score ranges between 13 and 91 points,
Sense of coherence (SOC) | Change from base-line scores SOC-13 scale at 6 months
  What is the effect of interactive patient education in supervised study groups on the participants' sense of coherence (measured by changes in scores in SOC-13 scale in Swedish9 from baseline to 6 months after baseline). Antonovsky developed the 29 item Orientation to Life Questionnaire to measure the sense of coherence, having 11 items measuring comprehensibility, 10 items measuring manageability, and 8 items measuring meaningfulness. The response alternatives are a semantic scale of 1 point to 7 points. The questionnaire yields a summed score with a range from 29 to 203. A shorter version of 13 questions of the original form was developed by Antonovsky, where the score ranges between 13 and 91 points,
Sense of coherence (SOC) | Change from base-line scores SOC-13 scale at 12 months
  What is the effect of interactive patient education in supervised study groups on the participants' sense of coherence (measured by changes in scores in SOC-13 scale in Swedish9 from baseline to 12 months after baseline). Antonovsky developed the 29 item Orientation to Life Questionnaire to measure the sense of coherence, having 11 items measuring comprehensibility, 10 items measuring manageability, and 8 items measuring meaningfulness. The response alternatives are a semantic scale of 1 point to 7 points. The questionnaire yields a summed score with a range from 29 to 203. A shorter version of 13 questions of the original form was developed by Antonovsky, where the score ranges between 13 and 91 points,
Health literacy | Change from base-line scores HLS-EU-Q16-SE scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' health literacy (measured by change in scores in HLS-EU-Q16-SE from baseline to 3 months after baseline). The instrument consists of 16 items focusing on four HL dimensions reflecting perceived ease or difficulty in an individual's ability to access/obtain health information, understand health information (not only in written form), process/appraise health information, and apply/use health information. More specifically, the 16 items include perceived skills for understanding health information, where to seek consultation and health information on prevention, early detection, and health care, health warnings, advice given by family and friends, how to seek a second opinion, and how to apply advice given by care providers. Response options include "very easy," "easy," "difficult," and "very difficult."
Health literacy | Change from base-line scores HLS-EU-Q16-SE scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' health literacy (measured by change in scores in HLS-EU-Q16-SE from baseline to 6 months after baseline). The instrument consists of 16 items focusing on four HL dimensions reflecting perceived ease or difficulty in an individual's ability to access/obtain health information, understand health information (not only in written form), process/appraise health information, and apply/use health information. More specifically, the 16 items include perceived skills for understanding health information, where to seek consultation and health information on prevention, early detection, and health care, health warnings, advice given by family and friends, how to seek a second opinion, and how to apply advice given by care providers. Response options include "very easy," "easy," "difficult," and "very difficult."
Health literacy | Change from base-line scores HLS-EU-Q16-SE scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' health literacy (measured by change in scores in HLS-EU-Q16-SE from baseline to 12 months after baseline). The instrument consists of 16 items focusing on four HL dimensions reflecting perceived ease or difficulty in an individual's ability to access/obtain health information, understand health information (not only in written form), process/appraise health information, and apply/use health information. More specifically, the 16 items include perceived skills for understanding health information, where to seek consultation and health information on prevention, early detection, and health care, health warnings, advice given by family and friends, how to seek a second opinion, and how to apply advice given by care providers. Response options include "very easy," "easy," "difficult," and "very difficult."
General self-efficacy | Change from base-line scores S-GSE scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' general self-efficacy (measured as change in scores in S-GSE from baseline to 3 months after baseline). About: This scale is a self-report measure of self-efficacy.
  Items: 10 Reliability:
  Internal reliability for GSE = Cronbach's alphas between .76 and .90
  Validity:
  The General Self-Efficacy Scale is correlated to emotion, optimism, work satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety.
  Scoring:
  All questions 1 2 3 4 The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General self-efficacy | Change from base-line scores S-GSE scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' general self-efficacy (measured as change in scores in S-GSE from baseline to 6 months after baseline). About: This scale is a self-report measure of self-efficacy.
  Items: 10 Reliability:
  Internal reliability for GSE = Cronbach's alphas between .76 and .90
  Validity:
  The General Self-Efficacy Scale is correlated to emotion, optimism, work satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety.
  Scoring:
  All questions 1 2 3 4 The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General self-efficacy | Change from base-line scores S-GSE scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' general self-efficacy (measured as change in scores in S-GSE from baseline to 12 months after baseline). About: This scale is a self-report measure of self-efficacy.
  Items: 10 Reliability:
  Internal reliability for GSE = Cronbach's alphas between .76 and .90
  Validity:
  The General Self-Efficacy Scale is correlated to emotion, optimism, work satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety.
  Scoring:
  All questions 1 2 3 4 The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Social function | Change from base-line scores sub scale "Social function" of RAND-36 at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' social function (measured as change in scores in the two questions used in the sub scale "Social function" of RAND-36 from baseline to 3 months after baseline). The RAND 36-Item Health Survey laps eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key. Note that all items are scored so that a high score defines a more favourable health state.
Social function | Change from base-line scores sub scale "Social function" of RAND-36 at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' social function (measured as change in scores in the two questions used in the sub scale "Social function" of RAND-36 from baseline to 6 months after baseline). The RAND 36-Item Health Survey (Version 1.0) laps eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key given. Note that all items are scored so that a high score defines a more favourable health state. I
Social function | Change from base-line scores sub scale "Social function" of RAND-36 at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' social function (measured as change in scores in the two questions used in the sub scale "Social function" of RAND-36 from baseline to 12 months after baseline). The RAND 36-Item Health Survey (Version 1.0) laps eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key given. Note that all items are scored so that a high score defines a more favourable health state.
Work ability | Change from base-line scores WAI scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' work ability (measured as change in scores in WAI from baseline to 3 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Work ability | Change from base-line scores WAI scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' work ability (measured as change in scores in WAI from baseline to 6 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Work ability | Change from base-line scores WAI scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' work ability (measured as change in scores in WAI from baseline to 12 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Job content | Change from base-line scores Karasek Job Content Questionnaire scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' job content (measured as change in score in Karasek Job Content Questionnaire from baseline to 3 months after baseline). Designed to measure scales assessing psychological demands, decision latitude, social support, physical demands, and job insecurity.
Job content | Change from base-line scores Karasek Job Content Questionnaire scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' job content (measured as change in score in Karasek Job Content Questionnaire from baseline to 6 months after baseline). Designed to measure scales assessing psychological demands, decision latitude, social support, physical demands, and job insecurity.
Job content | Change from base-line scores Karasek Job Content Questionnaire scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' job content (measured as change in score in Karasek Job Content Questionnaire from baseline to 12 months after baseline). Designed to measure scales assessing psychological demands, decision latitude, social support, physical demands, and job insecurity.
Total number of net and gross sick leave days | Change from base-line total number of net and gross sick leave days at 3 months
  What is the effect of interactive patient education in supervised study groups on the total number of net and gross sick leave days during the follow-up period (measured as change in measures defined by the Swedish Social Insurance Agency from baseline to 3 months after baseline).
Total number of net and gross sick leave days | Change from base-line total number of net and gross sick leave days at 6 months
  What is the effect of interactive patient education in supervised study groups on the total number of net and gross sick leave days during the follow-up period (measured as change in measures defined by the Swedish Social Insurance Agency from baseline to 6 months after baseline).
Total number of net and gross sick leave days | Change from base-line total number of net and gross sick leave days at 12 months
  What is the effect of interactive patient education in supervised study groups on the total number of net and gross sick leave days during the follow-up period (measured as change in measures defined by the Swedish Social Insurance Agency from baseline to 12 months after baseline).
Physical activity | Change from base-line scores LTPA (level of physical activity) scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' level of physical activity (measured as change in time spent on physical activities during leisure time according to LTPAI from baseline to 3 months after baseline).
Physical activity | Change from base-line scores LTPAI (level of physical activity) scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' level of physical activity (measured as change in time spent on physical activities during leisure time according to LTPAI from baseline to 6 months after baseline).
Physical activity | Change from base-line scores LTPAI (level of physical activity) scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' level of physical activity (measured as change in time spent on physical activities during leisure time according to LTPAI from baseline to 12 months after baseline).
BMI | Change from base-line scores BMI at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' Body Mass Index, BMI (measured as change in BMI from baseline to 3 months after baseline).
BMI | Change from base-line scores BMI at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' Body Mass Index, BMI (measured as change in BMI from baseline to 6 months after baseline).
BMI | Change from base-line scores BMI at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' Body Mass Index, BMI (measured as change in BMI from baseline to 12 months after baseline).
Symptoms of depression | Change from base-line scores MADRS-S scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of depression (measured as change in score in MADRS-S from baseline to 3 months after baseline).
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Symptoms of depression | Change from base-line scores MADRS-S scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of depression (measured as change in score in MADRS-S from baseline to 6 months after baseline).
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Symptoms of depression | Change from base-line scores MADRS-S scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of depression (measured as change in score in MADRS-S from baseline to 12 months after baseline).
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Symptoms of anxiety | Change from base-line scores GAD-7 scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of anxiety (measured change in score in GAD-7 from baseline to 3 months after baseline).
  Management Scores ≥10: Further assessment (including diagnostic interview and mental status examination) and/or referral to a mental health professional recommended.
  Score Symptom Severity Comments 5-9 Mild Monitor 10*-14 Moderate Possible clinically significant condition >15 Severe Active treatment probably warranted
Symptoms of anxiety | Change from base-line scores GAD-7 scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of anxiety (measured change in score in GAD-7 from baseline to 6 months after baseline).
  Score Symptom Severity Comments 5-9 Mild Monitor 10*-14 Moderate Possible clinically significant condition >15 Severe Active treatment probably warranted
Symptoms of anxiety | Change from base-line scores GAD-7 scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of anxiety (measured change in score in GAD-7 from baseline to 12 months after baseline).
  Score Symptom Severity Comments 5-9 Mild Monitor 10*-14 Moderate Possible clinically significant condition >15 Severe Active treatment probably warranted
Symptoms of exhaustion | Change from base-line scores KEDS scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of exhaustion (measured as change in score in KEDS from baseline to 3 months after baseline). items
  9 items/symptoms Scoring 0-6/item Total 0-54
  =/>19 p exhaustion
Symptoms of exhaustion | Change from base-line scores KEDS scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of exhaustion (measured as change in score in KEDS from baseline to 6 months after baseline).
  9 items/symptoms Scoring 0-6/item Total 0-54
  =/>19 p exhaustion
Symptoms of exhaustion | Change from base-line scores KEDS scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participants' symptoms of exhaustion (measured as change in score in KEDS from baseline to 12 months after baseline).
  9 items/symptoms Scoring 0-6/item Total 0-54
  =/>19 p exhaustion
Pain catastrophizing | Change from base-line scores pain catastrophizing scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participant pain catastrophizing (measured as change in score in PCS from baseline to 3 months after baseline).
  13 items Degree 0 - not at all
  1. - to a slight degree
  2. - to a moderate degree
  3. - to a great degree
  4. - all the time
Pain catastrophizing | Change from base-line scores pain catastrophizing scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participant pain catastrophizing (measured as change in score in PCS from baseline to 6 months after baseline).
  13 items Degree 0 - not at all
  1. - to a slight degree
  2. - to a moderate degree
  3. - to a great degree
  4. - all the time
Pain catastrophizing | Change from base-line scores pain catastrophizing scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participant pain catastrophizing (measured as change in score in PCS from baseline to 12 months after baseline).
  13 items Degree 0 - not at all
  1. - to a slight degree
  2. - to a moderate degree
  3. - to a great degree
  4. - all the time
Participant pain | Change from base-line scores OMPSQ scale at 3 months
  What is the effect of interactive patient education in supervised study groups on participant pain (measured as change in score in OMPSQ from baseline to 3 months after baseline). A higher score indicates a higher disability. Maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Participant pain | Change from base-line scores OMPSQ scale at 6 months
  What is the effect of interactive patient education in supervised study groups on participant pain (measured as change in score in OMPSQ from baseline to 6 months after baseline).
  Maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Participant pain | Change from base-line scores OMPSQ scale at 12 months
  What is the effect of interactive patient education in supervised study groups on participant pain (measured as change in score in OMPSQ from baseline to 12 months after baseline).
  Maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Pain spreading | Change from base-line scores in number of painful body regions at 3 months
  What is the effect of interactive patient education in supervised study groups on participant pain spreading (measured as change in number of painful body regions from baseline to 3 months after baseline). The diagram documents pain in 19 anatomic areas. Based on the distribution of the anatomic areas, we established six different body regions. Generalized linear regression was used to evaluate the association between the number of painful nonindex body regions (categorized as 0; 1-2; or 3-6) with our measures of interest. Participants reporting no body pain, low (1-2 regions) and high (≥ 3 regions).
Pain spreading | Change from base-line scores in number of painful body regions at 6 months
  What is the effect of interactive patient education in supervised study groups on participant pain spreading (measured as change in number of painful body regions from baseline to 6 months after baseline). The diagram documents pain in 19 anatomic areas. Based on the distribution of the anatomic areas, we established six different body regions. Generalized linear regression was used to evaluate the association between the number of painful nonindex body regions (categorized as 0; 1-2; or 3-6) with our measures of interest. Participants reporting no body pain, low (1-2 regions) and high (≥ 3 regions).
Pain spreading | Change from base-line scores in number of painful body regions at 12 months
  What is the effect of interactive patient education in supervised study groups on participant pain spreading (measured as change in number of painful body regions from baseline to 12 months after baseline). The diagram documents pain in 19 anatomic areas. Based on the distribution of the anatomic areas, we established six different body regions. Generalized linear regression was used to evaluate the association between the number of painful nonindex body regions (categorized as 0; 1-2; or 3-6) with our measures of interest. Participants reporting no body pain, low (1-2 regions) and high (≥ 3 regions).
Trust in own know-how | Change from base-line scores in questions about trust in own know-how and ability to improving health at 3 months
  What is the effect of interactive patient education in supervised study groups on participant trust in own know-how and ability related to improving health (measured as change in score in questions about trust in own know-how and ability to improving health from baseline to 3 months after baseline).
Trust in own know-how | Change from base-line scores in questions about trust in own know-how and ability to improving health at 6 months
  What is the effect of interactive patient education in supervised study groups on participant trust in own know-how and ability related to improving health (measured as change in score in questions about trust in own know-how and ability to improving health from baseline to 6 months after baseline).
Trust in own know-how | Change from base-line scores in questions about trust in own know-how and ability to improving health at 12 months
  What is the effect of interactive patient education in supervised study groups on participant trust in own know-how and ability related to improving health (measured as change in score in questions about trust in own know-how and ability to improving health from baseline to 12 months after baseline).
Partners in health care | Change from base-line scores in questions about informed as a patient and being a partner in health care at 3 months
  What is the effect of interactive patient education in supervised study groups on participants being informed as patients and being a partners in health care (measured as change in score in questions about informed as a patient and being a partner in health care from baseline to 3 months after baseline).
Partners in health care | Change from base-line scores in questions about informed as a patient and being a partner in health care at 6 months
  What is the effect of interactive patient education in supervised study groups on participants being informed as patients and being a partners in health care (measured as change in score in questions about informed as a patient and being a partner in health care from baseline to 6 months after baseline).
Partners in health care | Change from base-line scores in questions about informed as a patient and being a partner in health care at 12 months
  What is the effect of interactive patient education in supervised study groups on participants being informed as patients and being a partners in health care (measured as change in score in questions about informed as a patient and being a partner in health care from baseline to 12 months after baseline).
Visits to primary health care | Change from base-line proportion if they had to visit the primary health care center during the preceding two months, at 3 months
  What is the effect of interactive patient education in supervised study groups on participant visits to primary health care (research subjects are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 3 months. The measurement is the change in proportion of research subjects who visited the primary health care center).
Visits to primary health care | Change from base-line proportion if they had to visit the primary health care center during the preceding two months, at 6 months
  What is the effect of interactive patient education in supervised study groups on participant visits to primary health care (research subjects are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 6 months. The measurement is the change in proportion of research subjects who visited the primary health care center).
Visits to primary health care | Change from base-line proportion if they had to visit the primary health care center during the preceding two months, at 12 months
  What is the effect of interactive patient education in supervised study groups on participant visits to primary health care (research subjects are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 12 months. The measurement is the change in proportion of research subjects who visited the primary health care center).

CONTACTS AND LOCATIONS:
Locations (1):
- Dominique Hange, Gothenburg, Region Vastra Gotaland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lofgren M, Nordeman L, Ariai N, Bjorkelund C, Rembeck G, Svenningsson I, Tornbom K, Hange D. Effect on work ability and health-related quality of life following an interactive patient education aiming to increase sense of coherence and health literacy - the LEARN-to-COPE cluster randomized trial. Scand J Prim Health Care. 2025 Dec;43(4):805-820. doi: 10.1080/02813432.2025.2507859. Epub 2025 May 22. PMID 40405458

DOCUMENTS (1):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04254367/Prot_000.pdf